CLINICAL TRIAL: NCT04691700
Title: GOREISAN for Heart Failure (GOREISAN-HF) Trial
Acronym: GOREISAN-HF
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Professor of Medicine, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y0075; jRCT (Registry Identifier: jRCTs051200101)
Record Dates: First submitted 2020-12-20; First posted 2020-12-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Edema; Traditional Japanese Medicine; Kampo Medicine; Clinical Trial
Keywords: Heart Failure; Edema; Traditional Japanese Medicine; Goreisan (TJ-17); Clinical Trial
MeSH Terms: conditions — Heart Failure; Edema | interventions — oryeongsan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goreisan (Active Comparator): Goreisan (TJ-17) will be added at a dose of 7.5g per day to standard treatment
  Interventions: Drug: Goreisan
- No Goreisan (Active Comparator): Standard treatment without Goreisan (TJ-17)
  Interventions: Drug: Standard Treatment

INTERVENTIONS:
Drug: Goreisan — Add Goreisan 7.5g per day to standard treatment with the intention to reduce or discontinue the existing diuretics
  Arms: Goreisan
Drug: Standard Treatment — Standard therapy without Goreisan
  Arms: No Goreisan

SUMMARY:
The objective of the GOREISAN-HF trial is to assess the effect of the administration of Goreisan (TJ-17) plus standard therapy compared to standard therapy alone on the improvement rate of cardiac edema and clinical outcomes in worsening congestive heart failure with volume overload.

DETAILED DESCRIPTION:
Current guidelines recommend the use of loop diuretics as an indication for class I to improve HF symptoms regardless of left ventricular ejection fraction. Loop diuretics, however, are known to activate the renin-angiotensin-aldosterone system and the sympathetic nervous system, which could accelerate HF progression. Loop diuretics could also cause worsening renal function and electrolyte disturbance, and it is desirable to have an alternative drug to loop diuretics to effectively relieve congestive symptoms. Goreisan (TJ-17), a traditional Japanese medicine composed of five herbal medicines, has long been used in Japan to treat impairments of the regulation of body fluid homeostasis, including edema, and has been less likely to cause renal dysfunction and electrolyte abnormalities. We therefore planned a multicenter, randomized, interventional, parallel assignment, open-label treatment trial to evaluate the long-term effect of in-hospital initiation of Goreisan, when added to standard therapy, in patients with worsening congestive heart failure and clear signs of volume overload.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed congestive heart failure (CHF) by Framingham criteria
* CHF patients with cardiac edema and signs due to cardiac edema (signs of fluid overload: lower limb edema, pulmonary effusion, or pulmonary congestion on chest x-ray)
* Elevated N-terminal pro brain-type natriuretic peptide (NT-proBNP) ≥300 pg/mL or brain natriuretic peptide (BNP) ≥100 pg/mL at enrollment
* Patients ≥ 20 years of age, male or female
* Provision of signed informed consent before any assessment is performed

Exclusion Criteria:

* Valvular repair/replacement within 12 weeks prior to enrolment or planned to undergo any of these operations after randomization
* Implantation of a cardiac resynchronization therapy (CRT) within 12 weeks prior to enrollment or intent to implant a CRT device
* Previous cardiac transplantation or implantation of a ventricular assistance device or similar device, or implantation expected after randomization
* End-stage renal failure (estimated glomerular filtration rate [eGFR] <15 mL/min/1.73m2) at enrollment
* Patients who are expected to have a life expectancy of 6 months or less
* Acute coronary syndrome at screening
* Women of child-bearing potential or women who have a positive pregnancy test at enrolment or randomization
* Treatment with herbal medicine at enrollment
* Confirmed poor tolerability of Goreisan (including cinnamon allergy)
* Considered not appropriate for the participation of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1179 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of cardiac edema | 1 year
  Cardiac edema is defined as conditions having one or more following conditions: lower limb edema, pleural effusion, or pulmonary congestion on chest x-ray. Lower limb edema, pleural effusion, and pulmonary congestion are assessed by investigators. Improvement is defined as the disappearance of all signs of cardiac edema.
Composite endpoint of all-cause death or hospitalization | 3 years
  Composite of death from any cause or hospitalization from any cause.

SECONDARY OUTCOMES:
Change in the Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary score | 6 months
  The KCCQ is a validated self-administered instrument of quality of life and health status in heart failure (HF) patients. The clinical summary score is a composite assessment of physical limitation, total symptom score, health-related quality of life, and social limitation scores. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Change in loop diuretics dose | 6 months
  Loop diuretic dose will be calculated as furosemide-equivalent dose.
Change in loop diuretics dose | 1 year
  Loop diuretic dose will be calculated as furosemide-equivalent dose.
Composite endpoint of sustained decline in eGFR ≥50%, ESRD (end stage renal disease) or renal death | 3 years
  End Stage Renal Disease (ESRD) is defined as: Sustained eGFR <15 mL/min/1.73m2, Chronic dialysis treatment or, receiving a renal transplant. Renal death is defined as renal failure as the underlying cause of death.
Adverse drug event | 3 years
  Adverse drug event is an injury resulting from medical intervention related to any drug.
Change in a composite congestion score | 1 month
  Dyspnea, fatigue, orthopnea, jugular vein distention, rales, plueral effusion, and lower limb edema are assessed on a standardized 4-point scale ranging from 0 to 3. A composite congestion score is calculated by summing the individual scores for dyspnea, fatigue, orthopnea, jugular vein distention, rales, plueral effusion, and lower limb edema.
Change in a composite congestion score | 6 months
  Dyspnea, fatigue, orthopnea, jugular vein distention, rales, plueral effusion, and lower limb edema are assessed on a standardized 4-point scale ranging from 0 to 3. A composite congestion score is calculated by summing the individual scores for dyspnea, fatigue, orthopnea, jugular vein distention, rales, plueral effusion, and lower limb edema.
Change in a composite congestion score | 1 year
  Dyspnea, fatigue, orthopnea, jugular vein distention, rales, plueral effusion, and lower limb edema are assessed on a standardized 4-point scale ranging from 0 to 3. A composite congestion score is calculated by summing the individual scores for dyspnea, fatigue, orthopnea, jugular vein distention, rales, plueral effusion, and lower limb edema.
All-cause hospitalization | 3 years
  Hospitalization from any cause.
Composite endpoint of all-cause death or hospitalization for heart failure | 3 years
  Composite of death from any cause or hospitalization for heart failure.
Hospitalization for heart failure | 3 years
  Hospitalization for heart failure.
All-cause death | 3 years
  Death from any cause.
Non-cardiovascular death | 3 years
  Death other than death from cardiac or vascular diseases.
Change in New York Heart Association (NYHA) functional class | 6 months
  Change in New York Heart Association (NYHA) functional class, a well established grading scale to classify a patients' level of functionality based on the signs and symptoms of patient with heart failure.
Change in N-terminal pro brain-type natriuretic peptide (NT-proBNP) | 1 month
  Change in N-terminal pro brain-type natriuretic peptide (NT-proBNP).
Change in N-terminal pro brain-type natriuretic peptide (NT-proBNP) | 6 month
  Change in N-terminal pro brain-type natriuretic peptide (NT-proBNP).
Change in N-terminal pro brain-type natriuretic peptide (NT-proBNP) | 1 year
  Change in N-terminal pro brain-type natriuretic peptide (NT-proBNP).
Direct healthcare cost | 1 year
  Direct healthcare cost (Japanese Yen) from the time of randomization to 12 months was obained from the claim data patients.

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, PhD, Study Chair — Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Kyoto University Graduate School of Medicine, Kyoto, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yaku H, Kato T, Morimoto T, Kaneda K, Nishikawa R, Kitai T, Inuzuka Y, Tamaki Y, Yamazaki T, Kitamura J, Ezaki H, Nagao K, Yamamoto H, Isotani A, Takeshi A, Izumi C, Sato Y, Nakagawa Y, Matoba S, Sakata Y, Kuwahara K, Kimura T; GOREISAN-HF trial Investigators. Rationale and study design of the GOREISAN for heart failure (GOREISAN-HF) trial: A randomized clinical trial. Am Heart J. 2023 Jun;260:18-25. doi: 10.1016/j.ahj.2023.02.013. Epub 2023 Feb 24. PMID 36841318